CLINICAL TRIAL: NCT04852952
Title: Cross-cultural Translation of Oswestry Disability Index (ODI) Into Local Languages of Pakistan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/00931 Qandeel
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Descriptive analytical study to translate the Oswestry Disability Index into local languages of Pakistan that are, Pashto, Urdu, Punjabi, Sindhi, and Balochi languages. Along with validation of the translated versions by evaluating their validity and reliability in the people of Pakistan, speaking respective languages and suffering from low back pain. No such study has been previously conducted in the Pakistan region which translates the scale and follows the proper cross-cultural adaptation.

Condition or disease: Musculoskeletal disorders and disabilities caused by Low back pain, Non-probability Purposive Sampling would be used. The study will be conducted in relevant areas of Pakistan.

DETAILED DESCRIPTION:
As in the original study the main purpose of the Oswestry Disability Index is explained as to assess pain-related disability in persons with low back pain (LBP). The target population for the Oswestry are 3: acute, subacute, and chronic back pain client groups; with various conservative, surgical, and behavioural intervention groups.

The Oswestry Disability Index is one of the principal condition-specific outcome measures used for the investigation of low back musculoskeletal disorders. It is a self-administered questionnaire and consists of ten sections that are designed to assess the limitations of various daily life activities.

Each section is scored on a 0-5 scale, 5 is for maximum disability. The index is calculated by dividing the total score by the total possible score, which is multiplied by 100 and expressed as a percentage. Thus, for every unanswered question, the denominator is reduced by 5. If a patient marks two or more statements in a question, the highest-scoring statement is recorded as a true indication of disability. The questionnaire takes 3.5-5 min to complete andapproximately1 min to score.

At present worldwide there are a lot of health care workers who are using the Oswestry Disability Index for low back pain assessment and this scale is also providing good measurement but this scale is in the English language and there are a lot of people here in Pakistan who don't understand English. Pakistan is a country with different languages and cultures. The most commonly spoken and understood languages in Pakistan are Urdu the national language of Pakistan, Pashto, Punjabi, Sindhi, and Balochi. Therefore it is highly needed to translate this questioner into different languages so that the patient would be able to answer them easily according to their understanding. The validity and reliability of the translated versions will also be checked.

The translation and cultural adaptation processes would start after obtaining approval from the developer of the original Oswestry Disability Index scale. This would be done according to WHO guidelines. Translation will be done by symmetrical category. The purpose will be to gain uniformity in the translation of tool in both the Target language and Source language. This will involve 5 steps. (Forward translation, synthesis 1, Back translation, synthesis 2 and pilot testing.) Phase 2 would be done according to the standard guidelines in which psychometric properties will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patient both female and male having age group equal or >18.
* Patients should be capable to complete the questionnaire without any help.
* Diagnosed with nonspecific low back pain for more than 3 months.

Exclusion Criteria:

* Any serious conditions like neurological conditions which would not allow the patient to fill the questionnaire independently, any infection, tumour, spinal surgery, or any other rheumatological disease will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1000
Sampling Method: Non-Probability Sample
Enrollment: 576 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-12-23 (Estimated); Study Completion 2022-12-27 (Estimated)

PRIMARY OUTCOMES:
Oswestry disability Index translated versions | 1 year
  Self report versions. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

SECONDARY OUTCOMES:
Reliability of translated versions of Oswestry disability Index | 1 year
  To determine the reliability of cross-culturally adapted and the Oswestry disability Index translated versions in patients with the back pain of respective languages۔ Reliability or reproducibility refers to the ability of a measure to produce the same results when administered at two intervals between different visits of the patient. Thus this will be measured through test re-test reliability.
Validity of translated versions of Oswestry disability Index | 1 year
  To determine the validity of cross-culturally adapted and the translated Oswestry disability Index versions in patients with the back pain of respective languages۔ Validity is how accurate the results are. Thus this will be measured through various parameters to validate the translated versions as appropriate and applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joshi VD, Raiturker PP, Kulkarni AA. Validity and reliability of English and Marathi Oswestry Disability Index (version 2.1a) in Indian population. Spine (Phila Pa 1976). 2013 May 15;38(11):E662-8. doi: 10.1097/BRS.0b013e31828a34c3. PMID 23380824
- [Background] Yakut E, Duger T, Oksuz C, Yorukan S, Ureten K, Turan D, Frat T, Kiraz S, Krd N, Kayhan H, Yakut Y, Guler C. Validation of the Turkish version of the Oswestry Disability Index for patients with low back pain. Spine (Phila Pa 1976). 2004 Mar 1;29(5):581-5; discussion 585. doi: 10.1097/01.brs.0000113869.13209.03. PMID 15129077
- [Background] Mousavi SJ, Parnianpour M, Mehdian H, Montazeri A, Mobini B. The Oswestry Disability Index, the Roland-Morris Disability Questionnaire, and the Quebec Back Pain Disability Scale: translation and validation studies of the Iranian versions. Spine (Phila Pa 1976). 2006 Jun 15;31(14):E454-9. doi: 10.1097/01.brs.0000222141.61424.f7. PMID 16778675
- See also: Development of Brazilian version of ODI scale — https://pubmed.ncbi.nlm.nih.gov/17304141/